### INFORMED CONSENT FORM

in relation to the research project: "Fostering Ukraine's capacity in delivery and research of innovative evidence-based PTSD treatment (Lux4UA)"

| I,, | have read and understood the information |
|---|---|
| sheet regarding the above-mentioned research project | (Lux4UA Project) conducted by the research |
| team from the University of Luxembourg (UNILU), th | e Centre of Mental Health and Rehabilitation |
| "Forest Glade" of the Ministry of Health of Ukraine (Re | CFG), the National Psychological Association |
| of Ukraine (NPAU). I have been informed orally and i | n writing about the nature, purpose, duration, |
| procedures, potential risks, and benefits of participatin | g in the Lux4UA Project, and I have had the |
| opportunity to ask questions. | |

I understand that the Lux4UA Project aims to evaluate the **effectiveness and feasibility of the Reconsolidation of Traumatic Memories (RTM) Protocol** for PTSD treatment in Ukraine. My participation involves receiving either the RTM Protocol or another recognised trauma-focused therapy (treatment-as-usual) and completing questionnaires before, after, and at follow-up stages (6 and 12 months after treatment) as part of this study. The collected data will include age, gender, trauma type, diagnosis and symptoms, therapy experience.

### I have been informed that:

- Participation is voluntary, and I can withdraw my consent at any time without giving a reason and without any consequences for my care, which will be replaced with evidence-based alternatives.
- My personal data will be processed according to the EU General Data Protection Regulation (GDPR) and the Law of Ukraine on the Protection of Personal Data.
- All my personal information will be anonymised for research purposes.
- No identifiable data will be shared beyond the project's authorised team members.
- I have the right to **withdraw from the study at any time**, without giving a reason and without any negative consequences.
- I may request the deletion of my data or object to its further processing by contacting the research team.

## Please indicate your consent below:

| Statement | Yes | No |
|---|---|---|
| I consent to participate in this research study, including receiving PTSD treatment and | and _ | |
| completing questionnaires. | | |
| I agree that my anonymised data can be used for scientific publications and policy | | $ \Box $ |
| recommendations. | Ш | Ш |
| I agree to complete satisfaction surveys at the end of the treatment. | | |
| I agree to participate in a follow-up contact at 6 and 12 months after the treatment. | | |
| I agree to the data I provide being archived and used in anonymised form for other | | |
| research in the metal health area beyond the Lux4UA Project. | | |
| I voluntarily agree to take part in the Lux4UA Project. | | |

### **PARTICIPANT**

| Last name: |
|---|
| First name: |
| Email-address |
| Phone number |
| Place & date: |
| Signature: |
| RESEARCH COORDINATOR I have explained the purpose, procedures, risks, and benefits of Lux4UA Project to the participant named above and answered all their questions. Last name: First name: Place & date: |
| Signature: |
| D. w. darked a construction |

# **D-related contacts:**

NPA Data Protection Officer (email: <a href="mailto:dpo@npa-ua.org">dpo@npa-ua.org</a>; address: 12 Kozhumiatska Street, 04071, Kyiv, Ukraine (Nadia Diatel)

RCFG Protection Officer (email: dataprotection.forestglade@mailbox.org; address: 25, Line 7, Puscha-Vodytsia, 04114, Kyiv, Ukraine (Marta Vulchyn)